CLINICAL TRIAL: NCT04154306
Title: Effects of Fermented Red Clover on Muscle Strength and Muscle Protein Signaling in Postmenopausal Women
Brief Title: Effects of Fermented Red Clover on Muscle Strength and Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Estrogen_2019
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2019-10

CONDITIONS: Estrogen Deficiency
Keywords: Isoflavones; Red clover; Muscle Function; Postmenopausal women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Red clover (Experimental)
  Interventions: Dietary Supplement: Red clover

INTERVENTIONS:
Dietary Supplement: Red clover — 2 weeks of Red clover
  Arms: Red clover
Dietary Supplement: Placebo — 2 weeks of Placebo
  Arms: Placebo

SUMMARY:
The project is designed as a randomized controlled, double-blinded, cross-over trial, including 10 healthy postmenopausal women consuming fermented red clover extract or placebo twice daily over a two-week period. After the first trial (two weeks), participants will undergo a two-week washout period, after which they will receive the opposite trial drink for two weeks. The trial period runs over six weeks. Before each of the two trial rounds, participants will meet in the laboratory and perform muscle strength tests (trial days 1 and 3). After each trial round (trial days 2 and 4), participants will meet fasting in the laboratory, and a blood test and a muscle biopsy will be taken initially. Next, the subject consumes the test drink (placebo or red clover extract) before the subject performs a strength training session with one leg. Right after the training session, the subject consumes a protein drink. Three hours after the protein drink, another muscle biopsy is taken. During the period from the protein drink to the final biopsy, the subject performs two muscle strength tests (respectively grip strength and maximum upper arm muscle strength (biceps)). The primary target parameter is muscle protein signaling measured in the muscle tissue samples using the western blotting method.

ELIGIBILITY:
Inclusion Criteria:

* maximum of 5 years since last menstrual bleeding
* Minimum of 6 months since last menstrual bleeding

Exclusion Criteria:

* Performed systematic resistance training within the last 6 months
* Smoker
* Using any form of medicine influencing the effects of resistance training

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein signalling measured by western blotting | Change from pre to 3 hours post training
  Change in protein content between two time points

SECONDARY OUTCOMES:
Forearm and biceps strength measured by maximal isometric muscle strength | Change from Pre to post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark